CLINICAL TRIAL: NCT02715869
Title: Impact of Variable Types of Preconditioning Upon the Inotrope Score in Adult Patients, Undergoing Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Lecturer of Anesthesia and critical care Medicine, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00009901
Record Dates: First submitted 2016-03-17; First posted 2016-03-22 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Myocardial Ischemia
Keywords: Myocardial Preconditioning, inotropic score
MeSH Terms: conditions — Myocardial Ischemia | interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A pharmacologic cardiac preconditioning (Active Comparator): Sevoflurane as a pharmacologic preconditioner for the heart
  Interventions: Drug: A pharmacologic cardiac preconditioning (Sevoflurane)
- B ischeamic preconditioning (Active Comparator): ischemic preconditioning by inflation the cuff of blood pressure
  Interventions: Procedure: B ischeamic preconditioning

INTERVENTIONS:
Drug: A pharmacologic cardiac preconditioning (Sevoflurane) — A Patients are anaesthetized by Sevoflurane more than 1 mac.
  Arms: A pharmacologic cardiac preconditioning
Procedure: B ischeamic preconditioning — B ischemic preconditioning will be done after induction and before cardiopulmonary bypass by inflation the cuff of blood pressure above 200mmhg in the lower limb every 5 min for 3cycles
  Arms: B ischeamic preconditioning

SUMMARY:
Preconditioning (PC) of the heart occurs when brief exposure to a stimulus protects the heart from subsequent ischemia. PC stimulus may be (ischemic ; pharmacologic or Physical).

DETAILED DESCRIPTION:
Preconditioning (PC) of the heart occurs when brief exposure to a stimulus protects the heart from subsequent ischemia. PC stimulus may be ( ischemic ; pharmacologic or Physical)

Pharmacological PC may be induced by variable agents e.g. (Sevoflurane ;isoflorane, opioids etc)

Ischemic PC includes local; remote and the idea is temporary interruption of blood supply to the organ so that liberation of protective mediators occurs. The liberated mediators have favorable effects not only upon the myocardium, but it extend to protect other organs against inflammatory activation; ischemia reperfusion injury

Inotropic score (IS) is already an evident predictor of postoperative cardiac morbidity and mortality

Aim of the work:

Is to validate the impact of Sevoflurane versus ischemic & Sevoflurane PC upon postoperative inotropic score in adult patient undergoing open heart surgery

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old
* American Society of Anesthesiologists physical status II and III
* Patients scheduled for open heart surgery

Exclusion Criteria:

* Emergency surgery
* Clinically significant kidney or liver disease
* Patients allergic to local anesthetic
* Patients with prolonged cardiopulmonary bypass time (>120 min)
* Patients required intra-aortic balloon pump
* Postoperative hemodynamic instability (including the occurrence of serious arrhythmia) or bleeding that required surgical re-exploration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-03; Primary Completion 2017-03 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Highest inotropic score | first 24 hour

CONTACTS AND LOCATIONS:
Overall Officials: Emad Zarief Kamel Said, M.D., Study Director — Department of Anesthesia, faculty of Medicine, Assiut University
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No